CLINICAL TRIAL: NCT02342067
Title: A Phase 1, Multiple-Dose, Open-Label, Randomized, Crossover Study in Healthy Subjects to Assess the Effect of Pioglitazone (PGZ) on the Pharmacokinetics (PK) of Cenicriviroc Mesylate (CVC) and the Effect of CVC on the PK of PGZ
Brief Title: Pharmacokinetic and Safety Study of Cenicriviroc and Pioglitazone, When Dosed Alone or in Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tobira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 652-1-122
Record Dates: First submitted 2015-01-12; First posted 2015-01-19 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
MeSH Terms: interventions — cenicriviroc; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Cenicriviroc, PGZ, CVC+PGZ) (Experimental): Treatment A: CVC 150 mg QD for 10 days followed by 10-day washout Treatment B: PGZ 45 mg QD for 10 days Treatment C: co-administration of PGZ 45 mg QD + CVC 150 mg QD for 10 days
  Interventions: Drug: Cenicriviroc
- Group 2 (Pioglitazone, CVC, CVC+PGZ) (Experimental): Treatment B: PGZ 45 mg QD for 10 days followed by 10-day washout Treatment A: CVC 150 mg QD for 10 days Treatment C: co-administration of CVC 150 mg QD + PGZ 45 mg QD for 10 days
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Cenicriviroc — CVC 150 mg QD on Days 1-10, washout on Days 11-20, PGZ 45 mg QD on Days 21-30, and CVC 150 mg QD + PGZ 45 mg QD on Days 31-40
  Other Names: CVC 150 mg
  Arms: Group 1 (Cenicriviroc, PGZ, CVC+PGZ)
Drug: Pioglitazone — PGZ 45 mg QD on Days 1-10, washout on Days 11-20, CVC 150 mg QD on Days 21-30, and CVC 150 mg QD + PGZ 45 mg QD on Days 31-40
  Other Names: PGZ 45 mg
  Arms: Group 2 (Pioglitazone, CVC, CVC+PGZ)

SUMMARY:
A single center, open-label, fixed sequence study to evaluate the pharmacokinetics (PK) of Cenicriviroc (CVC) administered with and without Pioglitazone (PGZ), and to evaluate the PK of PGZ administered with and without CVC.

DETAILED DESCRIPTION:
This is a open-label, fixed-sequence, 3-period study being conducted in a single center to evaluate the following:

* PK of CVC administered with and without PGZ
* PK of PGZ administered with and without CVC
* Safety of CVC administered with and without PGZ
* Tolerability of CVC administered with and without PGZ

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* BMI ≥ 18 and ≤ 35 kg/m2
* No clinically relevant abnormalities based on medical history, physical examination, clinical laboratory evaluations, and 12-lead ECG
* Agree to comply with the study procedures and restrictions

Exclusion Criteria:

* Any disease or condition that might affect drug absorption, metabolism, or excretion, or clinically significant conditions as determined by the investigator
* History of stomach or intestinal surgery, except for fully healed appendectomy and/or cholecystectomy
* Serum ALT, AST or bilirubin ≥ grade 1 (ALT and AST > ULN - 3.0 x ULN; bilirubin > ULN - 1.5 x ULN) at screening
* Positive for HIV, HBV or HCV infection
* Use of any prescription drugs or prohibited medications within 30 days from the first dose of the study medication
* Use of alcohol-containing or caffeine-containing foods or beverages within 72 hours prior to the first dose of study medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Assessment of CVC, as measured by Cmax, Cmin and AUC | Predose (0 hours), 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours postdose on Days 10, 30 and 40
  PK profile will be calculated based on CVC exposure. Trough (predose) CVC plasma samples will be obtained prior to dosing on Days 2-9, 22-29, and 32-39.
Pharmacokinetic Assessment of PGZ, as measured by Cmax, Cmin and AUC | Predose (0 hours), 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours postdose on Days 10, 30 and 40
  PK profile will be calculated based on PGZ exposure. Trough (predose) CVC plasma samples will be obtained prior to dosing on Days 2-9, 22-29, and 32-39.

SECONDARY OUTCOMES:
Evaluation of Adverse Events | 40 days
  Evaluate adverse events
Changes from Baseline in Clinical Laboratory Tests | 40 days
  Evaluate changes from baseline in clinical laboratory tests including serum chemistry (ALT, AST, BUN, cholesterol, glucose), hematology (hemoglobin, red blood cell count, white blood cell count and differential), urinalysis (pH, glucose, ketones, protein, urobilinogen)
Changes from Baseline in 12-lead ECGs | 40 days
  Evaluate changes from baseline in 12-lead ECGs
Changes from Baseline in Vital Signs | 40 days
  Evaluate changes from baseline in vital signs, including blood pressure and pulse rate
Changes from Baseline in Physical Examinations | 40 days
  Evaluate changes from baseline in physical examinations

CONTACTS AND LOCATIONS:
Locations (1):
- DaVita Clinical Research, Lakewood, Colorado, United States